

**Royal Papworth Hospital NHS Foundation Trust** 

Cambridge Biomedical Campus Papworth Road Cambridge CB2 0AY

Tel: 01223 638000 www.royalpapworth.nhs.uk

Centre Number: *If applicable*Study Number: P0XXXX

Patient Identification Number:

## **CONSENT FORM**

Version 4.0 dated 03/09/19

**Study title:** Measurement of mucus plugging with computer tomography before and following implementation of the AffloVest in adults with bronchiectasis – a feasibility study.

Study IRAS ID:257616

Local Investigator: Mrs Siobhan Singh

## Please initial box

| 1. I confirm that I have read and understood the information sheet dated 03/09/19 | |
|---|---|
| (version 4.0) for the above study. I have had the opportunity to consider the | |
| information, ask questions and have had these answered satisfactorily. | |
| 2. I understand that my participation is voluntary and that I am free to withdraw | |
| at any time without giving any reason, without my medical care or legal rights being | |
| affected. | |
| 3. I understand that relevant sections of my medical notes and data collected during | |
| the study may be looked at by individuals from the NHS Trust, where it is relevant to | ) |
| my taking part in this research. Whenever possible this information will be | |
| anonymised. I give permission for these individuals to have access to my records. | |

4. I understand that if I wish to keep the AffloVest at the end of the study, my name, phone number and address will be shared with International Biophysics Corporation

| for purposes of warranty and servicing of the AffloVest. I give permission for this | | |
|---|---|---|
| information to be shared to International Biophysics Corporation (who are based in | | |
| the US) for this purpose | | |
| 5. I agree to my GP being informed of my participation in the study. | | |
| 6. I agree to take part in the above study. | | |
| 7. I consent to be contacted if applicable for future related studies or data collection | | |
| or for my data to be used for long term follow up studies and am aware I can | | |
| withdraw this consent at any point. | | |
| Name of Patient (PRINT) | Date | Signature |
| Name of Patient (PRINT) | Date | Signature |
| Name of person taking consent (PRINT | ) Date | Signature |
| reame of person taking consent (French | ) Date | Olgitatare |
| When completed: 1 for participant; 1 for researcher site file; 1 (original) to be kept in | | |
| medical notes. | | , |